CLINICAL TRIAL: NCT05409898
Title: Screening for Masked Hypertension in Young and Middle-aged Adults With Smart Wearable Devices (SMART)
Brief Title: Screening for Masked Hypertension With Smart Wearable Devices (SMART)
Acronym: SMART
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jing Liu (Other)
Collaborators: HUAWEI (Unknown)
Responsible Party: Sponsor-Investigator, Jing Liu, Director of the Department of Hypertension, Peking University People's Hospital
Organization: Peking University People's Hospital (Other)
Other Study IDs: 2022PHB108
Record Dates: First submitted 2022-06-03; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-06

CONDITIONS: Masked Hypertension
Keywords: asked hypertension, Smart wearable device
MeSH Terms: conditions — Masked Hypertension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: smart wearable device — screening masked hypertension with smart wearable devices

SUMMARY:
In recent years, a large number of consumer-grade and Smart Wearable Devices (SWD) such as smart watches, with BP measurement property, have entered the market and have a high configuration and utilization among young and middle-aged populations, but most of them are uncalibrated and have poor accuracy. Recently, several medical-grade smart BP watches have passed the national medical device registration test, which will provide an important tool for accurate screening of hypertension, especially masked hypertension, in young and middle-aged people.

"Screening for masked hypertension in young and middle-aged adults with smart wearable devices" （SMART）aims to screen for masked hypertension using smart BP watches that have been tested for national medical device registration. It is planned to include 200 young and middle-aged subjects with normal blood pressure (BP) in the clinic, who will wear the smart BP watch for 7 consecutive days (BP will be measured at least once in the morning and once in the evening, 2-3 times each time), and if the mean BP is >= 135/85 mmHg, it will be determined to be MK and recommended for further consultation and treatment.

DETAILED DESCRIPTION:
Masked hypertension (MH) is defined as elevated ambulatory or home blood pressure (BP), but normal office BP, often complicated with severe cardiovascular and renal damage. MH is easily missed and needs to be identified by "out-of-office" BP measurements such as ambulatory BP monitoring (ABPM) or home BP monitoring (HBPM). However, in clinical practice, ABPM has poor accessibility, high cost, and requires appointments, making it difficult to meet the demand; HBPM has better accessibility, but low utilization and irregular use are more prominent. In addition, these devices interfere with sleep and activity when measuring BP, so their clinical application is somewhat limited.

Smart wearable devices (SWD) can sense and record various physiological parameters of human body, and analyze the health status of individuals with the support of software algorithms. In recent years, a large number of consumer-grade and SWD such as smart watches, with BP measurement property, have entered the market and have a high configuration and utilization among young and middle-aged populations, but most of them are uncalibrated and have poor accuracy. Recently, several medical-grade smart BP watches have passed the national medical device registration test, which will provide an important tool for accurate screening of hypertension, especially MH, in young and middle-aged people.

"Screening for masked hypertension in young and middle-aged adults with smart wearable devices" （SMART） aims to screen for MH using smart BP watches that have been tested for national medical device registration. It is planned to include 200 young and middle-aged subjects with normal blood pressure in the clinic, who will wear the smart BP watch for 7 consecutive days (BP will be measured at least once in the morning and once in the evening, 2-3 times each time), and if the mean BP is >= 135/85 mmHg, it will be determined to be MK and recommended for further consultation and treatment.

ELIGIBILITY:
Inclusion Criteria:

1. 18-50 years of age, male or female
2. No clear previous history of hypertension and other cardiovascular diseases
3. Signed informed consent form

Exclusion Criteria:

1. Patients with established hypertension
2. History of severe heart, liver, or kidney disease
3. Inability to cooperate in completing the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will be recruited in the hospital in the volunteers who are interested in this project or those who are concern of the hypertension despite with norm tension during usual physical examinations.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-07 (Estimated); Primary Completion 2024-06 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Prevalence of masked hypertension | 7 days
  Average systolic/diastolic BP during 7 days of the observation period will be calculated.
  Office BP should be measured when the average BP is ≥135/85 mmHg during 7 days of continuous self-monitoring. If the office BP is < 140/90 mmHg at visit, "Masked Hypertension" will be diagnosed.
  The prevalence of masked hypertension will be calculated as the following:
  number of masked hypertension/number of subjects included.

SECONDARY OUTCOMES:
Prevalence of hypertension | 7 days
  Average systolic/diastolic BP during 7 days of the observation period will be calculated.
  Office BP should be measured when the average BP is ≥135/85 mmHg during 7 days of continuous self-monitoring. If the office BP is ≥140/90 mmHg at visit, the diagnosis will be "Hypertension".
  The prevalence of hypertension will be calculated as the following:
  number of hypertension/number of subjects included.

CONTACTS AND LOCATIONS:
Overall Officials: Jing Liu, MD, Study Chair — Peking University People's Hospital
Locations (1):
- Peking University People's Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No